CLINICAL TRIAL: NCT02887443
Title: An Open-label Study to Assess the Potential for Pre-systemic Inhibition of Cytochrome P450 3A4 (CYP3A) by Idebenone in Healthy Male Subjects Using Midazolam as a Substrate
Brief Title: A Study to Assess the Potential for Pre-systemic Inhibition of CYP3A by Idebenone Using Midazolam as a Substrate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SNT-I-017
Record Dates: First submitted 2016-08-03; First posted 2016-09-02 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Drug-Drug Interaction
MeSH Terms: interventions — idebenone

INTERVENTIONS:
Drug: Raxone (idebenone 150 mg) — Raxone (idebenone 300 mg t.i.d.) on days 3 and days 5 to 10
Drug: Midazolam 2,5 mg — Midazolam (2,5 mg single oral dose) on days 1, 3 and 10

SUMMARY:
This phase I open label study is conducted to assess the potential pharmacokinetic interaction of Raxone® with midazolam in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male aged 18 to 55 years.
2. A Body Mass Index (BMI) of 18-30. BMI = Body weight (kg) / Height (m)2.
3. Male subject willing to use an acceptable effective contraceptive measure for the entire duration of study participation.
4. No clinically significant abnormal serum biochemistry, haematology and urine examination values.
5. A negative urinary test for drugs of abuse and alcohol breath screen. A positive alcohol test may be repeated at the discretion of the Investigator.
6. Negative HIV and Hepatitis B and C results.
7. No clinically significant abnormalities in 12 lead electrocardiogram (ECG).
8. No clinically significant abnormalities in blood pressure, pulse or oral temperature.
9. No allergy or sensitivity to midazolam, idebenone or any of their excipients.
10. No current or past medical condition that might significantly affect the pharmacokinetic or pharmacodynamic response to midazolam.
11. Subject must be available to complete the study (including follow-up visit).
12. Subject must satisfy a medical examiner about their fitness to participate in the study.
13. Subject must provide written informed consent to participate in the study.
14. Covered by Health Insurance System and/or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

1. A clinically significant history of gastrointestinal disorder likely to influence drug absorption.
2. Use of any medication (prescription or OTC, including health supplements and herbal remedies, except paracetamol, within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose of trial medication.
3. Use of any medication known to induce or inhibit any of the enzymes within the CYP3A system within 28 days of Day 1, or grapefruit within 7 days of Day 1
4. Evidence of renal, hepatic dysfunction, cardiovascular or metabolic dysfunction.
5. History of obstructive sleep apnoea syndrome.
6. History of any significant drug allergy including benzodiazepine.
7. A clinically significant history of drug or alcohol abuse.
8. Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
9. Participation in a clinical trial of a New Chemical Entity within the previous 3 months or of a Marketed Product within the previous 30 days (or 5 times the half-life, whichever is longer).
10. Donation of 450 mL or more blood within the previous 3 months.
11. Smoking or use of tobacco products or substitutes within the previous 6 months, as determined at the Screening visit.
12. Need for administrative or legal supervision.
13. Subject who would receive more than 4500 euros as indemnities for participation in biomedical research within 12 months, including the indemnities for the present study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) from the time of dosing to the time of the last observed concentration (AUC0-t) | 13 days
Area Under the Curve (AUC) extrapolated to infinity from dosing time, based on the last observed concentration (AUC0-∞) | 13 days
Maximum plasma concentration (Cmax) | 13 days
Time to Maximum plasma concentration (Cmax) during a dosing interval (tmax) | 13 days
Terminal elimination half-life (t1/2) | 13 days
Clearance, calculated as dose/AUC0-∞ (CL/F) | 13 days
Volume of distribution during terminal phase after non-intravenous administration (Vz/F) | 13 days

SECONDARY OUTCOMES:
Area Under the Curve (AUC) from the time of dosing to the time of the last observed concentration (AUC0-t) | 13 days
Area Under the Curve (AUC) extrapolated to infinity from dosing time, based on the last observed concentration (AUC0-∞) | 13 days
Maximum plasma concentration (Cmax) | 13 days
Time to Maximum plasma concentration (Cmax) during a dosing interval (tmax) | 13 days
Terminal elimination half-life (t1/2) | 13 days
Clearance (CL) | 13 days
Clearance, calculated as dose/AUC0-∞ (CL/F) | 13 days
Volume of distribution (Vz) | 13 days
Volume of distribution during terminal phase after non-intravenous administration (Vz/F) | 13 days

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Optimed, Gières, France